CLINICAL TRIAL: NCT01834261
Title: Computational Modeling of Oxytocin in the Regulation of Trust
Brief Title: Brain Dynamics of Oxytocin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: Martinos Center for Biomedical Imaging (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 293408; N000141210393 (Other Grant/Funding Number: ONR)
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-01

CONDITIONS: Brain Dynamics in Healthy Adults
Keywords: oxytocin; trust; kinship; kin selection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin (Active Comparator): Healthy adult subjects will receive several puffs of Syntocinon Nasal Spray, 40IU, once, prior to MRI and/or MEG scanning.
  Interventions: Drug: Syntocinon Nasal Spray, 40IU; Drug: Syntocinon Placebo Formulation, 40IU
- Placebo (Placebo Comparator): Healthy adult subjects will receive several puffs of Syntocinon Placebo Formulation, 40IU, once, prior to MRI and/or MEG scanning.
  Interventions: Drug: Syntocinon Nasal Spray, 40IU; Drug: Syntocinon Placebo Formulation, 40IU

INTERVENTIONS:
Drug: Syntocinon Nasal Spray, 40IU — Subjects will be scanned twice. Prior to first brain scanning session, they will be randomly assigned to receive either Syntocinon or Placebo. Prior to second scanning session, they will receive what they have not received in the first session; i.e., same subjects will be receiving both Syntocinon and placebo on two different days.
Drug: Syntocinon Placebo Formulation, 40IU — Subjects will be scanned twice. Prior to first brain scanning session, they will be randomly assigned to receive either Syntocinon or Placebo. Prior to second scanning session, they will receive what they have not received in the first session; i.e., same subjects will be receiving both Syntocinon and placebo on two different days.

SUMMARY:
Oxytocin is a neuropeptide that is well known for its role in social and affiliative behavior in humans. Oxytocin receptors are significantly lowered in autistic individuals and administration of oxytocin has shown benefits in enhancing social recognition and behavior in autistic children. However, more recent research has refined the behavioral effects of oxytocin, moving away from the notion that the neuropeptide blindly induces love and trust, towards the view that it actually increases social perception in assessing friend vs. foe: supporting cohesion with 'insiders' and distrust and aggression for 'outsiders.' Oxytocin is responsible for the selective aggression shown by lactating female mammals protecting their young, an effect demonstrated also in humans, and has been shown to strengthen feelings of ethnocentrism. However, no neuroimaging study to date has investigated this effect, with the consequence that its neurobiological basis is still unknown.

The general aim of our study is to determine meso-circuit brain dynamics that underlie oxytocin's amplification of both trust and aggression; and specifically, using neuroimaging (fMRI, magnetoencephalography, and behavioral testing) whether oxytocin amplifies kinship bias by attenuating social reward learning.

DETAILED DESCRIPTION:
The purpose of the study is to understand how oxytocin affects brain and behavior. The study will compare Syntocinon Nasal Spray to placebo. The specific aims are to:

1. Determine the default circuitry of oxytocin (OT).
2. Determine time-course and gender differences for default neural response to OT.
3. Using an iterative version of the classical neuroeconomic game (Trust Study), behaviorally test whether OT down-regulates reward learning, thereby enhancing the effects of kinship bias, to account for the polarizing effects (in which OT increases trust for 'in-groups' and increases aggression for 'out-groups').
4. Identify the down-regulation of reward learning neurobiologically, via data-driven control systems modeling of the reward circuit using MRI (fMRI: time-series analysis of the orbitofrontal cortex, amygdala, anterior and posterior cingulate, and nucleus accumbens, and magnetic resonance spectroscopy: focusing on gamma-Aminobutyric acid neurotransmitters within the nucleus accumbens) and magnetoencephalography (focusing on the dynamics within the prefrontal cortex). FMRI and MRS will be conducted during the same MRI scan, while MEG will be conducted separately.

STUDY PROCEDURES:

Nasal Obstruction/Anosmia Screening: All potential subjects will be screened for total or partial anosmia and nasal congestion using the University of Pennsylvania Smell Identification Test (Psychological Assessment Resources, Lutz FL).

Pregnancy and Lactation Screening: Oxytocin is often used clinically to trigger labor in late-stage pregnancy. Although none of our subjects will be in late-stage pregnancy and subjects will be receiving dosages far smaller that those used to trigger labor, to be safe all potential female subjects will be urine screened for pregnancy immediately during the history and physical. Lactation screening will be performed via self-report, and is conducted to avoid confounds due to endogenously produced OT during the milk-ejection reflex.

Oxytocin/Placebo Procedures: Oxytocin intranasal spray is manufactured as the Syntocinon Nasal Spray. The typical dose oxytocin of for short-term intranasal use is 40IU, and has an expected half-life of 20 minutes. Placebos, identical in preparation except for the oxytocin component, will be administered in the same manner in a double blind procedure. To avoid bleed-through between conditions while controlling for order effects, sessions will not be mixed between drug and placebo conditions: each session, conducted on separate days, will be either 'drug' or 'placebo.'

Scanning Procedures: Scanning procedure for MRI will include: structural scan (6 minutes), fMRI or MRS resting state (10 minutes), and a neuroeconomic task scan (10 minutes). Scanning procedure for MEG will include: resting state (10 minutes), and a neuroeconomic task scan (20 minutes).

Behavioral Task: During scans, subjects will participate in an interactive neuroeconomic game, an iterative version of the classical "Trust Study". During this game, the subject ('investor') is first provided a sum of money. He then has the choice in terms of how much to invest in a fictional computer-generated trustee or, in forced-choice versions, to choose between different trustees. The trustee then sends some percentage back to the subject ('investor'), and the game iterates over many trials. Previous research has shown that OT disrupts participant's use of the optimal solution, eliciting greater "trust" in the trustee than would be expected by Nash Equilibrium. To modulate reward learning, algorithms for trustee behavior will be modulated towards greater and lesser generosity. To modulate kinship bias, trustees will be represented on the screen using faces of greater and lesser similarity to that of the subject, created using MorphMan video-editing software (STOIK Imaging, Moscow Russia).

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age

Exclusion Criteria:

* any significant known medical condition, including mental disorders (confounds interpretation of brain activity)
* metal in the body or claustrophobia (contraindicated for fMRI)
* current use of any type of psychotropic medication (confounds interpretation of brain activity)
* body mass index of greater than 30 (to permit matched dosing across subjects)
* pregnancy (contraindicated for OT)
* breastfeeding (lactation endogenously triggers OT, which would not permit a placebo condition)
* smoking (affects use of nasal spray)
* use of drugs of abuse (confounds interpretation of brain activity)
* blood pressure above the normal range (140/90 mm Hg) or controlled with medication (may theoretically increase risk for OT side-effects)
* anosmia (affects use of nasal spray)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lilianne Mujica-Parodi, PhD, Principal Investigator — Stony Brook University
Locations (3):
- United States (3):
  - Martinos Imaging Center at the McGovern Institute for Brain Research at MIT, Cambridge, Massachusetts
  - Martinos Center for Biomedical Research, Building 149, 13th Street, Charlestown, Massachusetts
  - Bioengineering Building , Stony Brook University, Stony Brook, New York

REFERENCES:
- [Background] Averbeck BB. Oxytocin and the salience of social cues. Proc Natl Acad Sci U S A. 2010 May 18;107(20):9033-4. doi: 10.1073/pnas.1004892107. Epub 2010 May 6. No abstract available. PMID 20448196
- [Background] Insel TR. The challenge of translation in social neuroscience: a review of oxytocin, vasopressin, and affiliative behavior. Neuron. 2010 Mar 25;65(6):768-79. doi: 10.1016/j.neuron.2010.03.005. PMID 20346754
- [Background] Baumgartner T, Heinrichs M, Vonlanthen A, Fischbacher U, Fehr E. Oxytocin shapes the neural circuitry of trust and trust adaptation in humans. Neuron. 2008 May 22;58(4):639-50. doi: 10.1016/j.neuron.2008.04.009. PMID 18498743
- [Background] Delgado MR. Fool me once, shame on you; fool me twice, shame on oxytocin. Neuron. 2008 May 22;58(4):470-1. doi: 10.1016/j.neuron.2008.05.005. PMID 18498730
- [Background] Kosfeld M, Heinrichs M, Zak PJ, Fischbacher U, Fehr E. Oxytocin increases trust in humans. Nature. 2005 Jun 2;435(7042):673-6. doi: 10.1038/nature03701. PMID 15931222
- [Background] Wermter AK, Kamp-Becker I, Hesse P, Schulte-Korne G, Strauch K, Remschmidt H. Evidence for the involvement of genetic variation in the oxytocin receptor gene (OXTR) in the etiology of autistic disorders on high-functioning level. Am J Med Genet B Neuropsychiatr Genet. 2010 Mar 5;153B(2):629-639. doi: 10.1002/ajmg.b.31032. PMID 19777562
- [Background] Park J, Willmott M, Vetuz G, Toye C, Kirley A, Hawi Z, Brookes KJ, Gill M, Kent L. Evidence that genetic variation in the oxytocin receptor (OXTR) gene influences social cognition in ADHD. Prog Neuropsychopharmacol Biol Psychiatry. 2010 May 30;34(4):697-702. doi: 10.1016/j.pnpbp.2010.03.029. Epub 2010 Mar 27. PMID 20347913
- [Background] Gregory SG, Connelly JJ, Towers AJ, Johnson J, Biscocho D, Markunas CA, Lintas C, Abramson RK, Wright HH, Ellis P, Langford CF, Worley G, Delong GR, Murphy SK, Cuccaro ML, Persico A, Pericak-Vance MA. Genomic and epigenetic evidence for oxytocin receptor deficiency in autism. BMC Med. 2009 Oct 22;7:62. doi: 10.1186/1741-7015-7-62. PMID 19845972
- [Background] Andari E, Duhamel JR, Zalla T, Herbrecht E, Leboyer M, Sirigu A. Promoting social behavior with oxytocin in high-functioning autism spectrum disorders. Proc Natl Acad Sci U S A. 2010 Mar 2;107(9):4389-94. doi: 10.1073/pnas.0910249107. Epub 2010 Feb 16. PMID 20160081
- [Background] Guastella AJ, Einfeld SL, Gray KM, Rinehart NJ, Tonge BJ, Lambert TJ, Hickie IB. Intranasal oxytocin improves emotion recognition for youth with autism spectrum disorders. Biol Psychiatry. 2010 Apr 1;67(7):692-4. doi: 10.1016/j.biopsych.2009.09.020. Epub 2009 Nov 7. PMID 19897177
- [Background] Rossignol DA. Novel and emerging treatments for autism spectrum disorders: a systematic review. Ann Clin Psychiatry. 2009 Oct-Dec;21(4):213-36. PMID 19917212
- [Background] Opar A. Search for potential autism treatments turns to 'trust hormone'. Nat Med. 2008 Apr;14(4):353. doi: 10.1038/nm0408-353. No abstract available. PMID 18391923
- [Background] Bartz J, Simeon D, Hamilton H, Kim S, Crystal S, Braun A, Vicens V, Hollander E. Oxytocin can hinder trust and cooperation in borderline personality disorder. Soc Cogn Affect Neurosci. 2011 Oct;6(5):556-63. doi: 10.1093/scan/nsq085. Epub 2010 Nov 29. PMID 21115541
- [Background] Bartz JA, Zaki J, Ochsner KN, Bolger N, Kolevzon A, Ludwig N, Lydon JE. Effects of oxytocin on recollections of maternal care and closeness. Proc Natl Acad Sci U S A. 2010 Dec 14;107(50):21371-5. doi: 10.1073/pnas.1012669107. Epub 2010 Nov 29. PMID 21115834
- [Background] Hahn-Holbrook J, Holt-Lunstad J, Holbrook C, Coyne SM, Lawson ET. Maternal defense: breast feeding increases aggression by reducing stress. Psychol Sci. 2011 Oct;22(10):1288-95. doi: 10.1177/0956797611420729. Epub 2011 Aug 26. PMID 21873570
- [Background] De Dreu CK, Greer LL, Van Kleef GA, Shalvi S, Handgraaf MJ. Oxytocin promotes human ethnocentrism. Proc Natl Acad Sci U S A. 2011 Jan 25;108(4):1262-6. doi: 10.1073/pnas.1015316108. Epub 2011 Jan 10. PMID 21220339
- [Background] Domes G, Lischke A, Berger C, Grossmann A, Hauenstein K, Heinrichs M, Herpertz SC. Effects of intranasal oxytocin on emotional face processing in women. Psychoneuroendocrinology. 2010 Jan;35(1):83-93. doi: 10.1016/j.psyneuen.2009.06.016. PMID 19632787
- [Background] Domes G, Heinrichs M, Glascher J, Buchel C, Braus DF, Herpertz SC. Oxytocin attenuates amygdala responses to emotional faces regardless of valence. Biol Psychiatry. 2007 Nov 15;62(10):1187-90. doi: 10.1016/j.biopsych.2007.03.025. Epub 2007 Jul 9. PMID 17617382
- [Background] Domes G, Heinrichs M, Michel A, Berger C, Herpertz SC. Oxytocin improves "mind-reading" in humans. Biol Psychiatry. 2007 Mar 15;61(6):731-3. doi: 10.1016/j.biopsych.2006.07.015. Epub 2006 Nov 29. PMID 17137561
- [Background] Dupont CP. Contact dermatitis in Dublin. Contact Dermatitis. 1979 Jan;5(1):61-2. doi: 10.1111/j.1600-0536.1979.tb05548.x. No abstract available. PMID 421469
- [Background] Kirsch P, Esslinger C, Chen Q, Mier D, Lis S, Siddhanti S, Gruppe H, Mattay VS, Gallhofer B, Meyer-Lindenberg A. Oxytocin modulates neural circuitry for social cognition and fear in humans. J Neurosci. 2005 Dec 7;25(49):11489-93. doi: 10.1523/JNEUROSCI.3984-05.2005. PMID 16339042
- [Background] Petrovic P, Kalisch R, Singer T, Dolan RJ. Oxytocin attenuates affective evaluations of conditioned faces and amygdala activity. J Neurosci. 2008 Jun 25;28(26):6607-15. doi: 10.1523/JNEUROSCI.4572-07.2008. PMID 18579733
- [Background] Pincus D, Kose S, Arana A, Johnson K, Morgan PS, Borckardt J, Herbsman T, Hardaway F, George MS, Panksepp J, Nahas Z. Inverse effects of oxytocin on attributing mental activity to others in depressed and healthy subjects: a double-blind placebo controlled FMRI study. Front Psychiatry. 2010 Oct 12;1:134. doi: 10.3389/fpsyt.2010.00134. eCollection 2010. PMID 21423444
- [Background] Singer T, Snozzi R, Bird G, Petrovic P, Silani G, Heinrichs M, Dolan RJ. Effects of oxytocin and prosocial behavior on brain responses to direct and vicariously experienced pain. Emotion. 2008 Dec;8(6):781-91. doi: 10.1037/a0014195. PMID 19102589
- [Background] MacDonald E, Dadds MR, Brennan JL, Williams K, Levy F, Cauchi AJ. A review of safety, side-effects and subjective reactions to intranasal oxytocin in human research. Psychoneuroendocrinology. 2011 Sep;36(8):1114-26. doi: 10.1016/j.psyneuen.2011.02.015. Epub 2011 Mar 23. PMID 21429671
- See also: Lab Website — http://www.lcneuro.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at MIT and at MGH (distinct populations of participants). They randomly received Syntocinon or Placebo (40 IU) first. 51 subjects consented. 10 dropped out prior to receiving either drug. 21 at MIT and 20 at MGH completed at least one visit where they received either placebo/oxytocin. A total of 39 completed both.
Pre-assignment Details: All subjects who consented and passed history and physical examination received both oxytocin and placebo on different days. Exclusion criteria included any significant known medical conditions, metal in the body or claustrophobia, current use of psychotropic medications, BMI > 30, pregnancy, breastfeeding, smoking, high blood pressure and anosmia.
Groups:
- Oxytocin, Then Placebo: Healthy adult subjects who received oxytocin before their first scan, and placebo before their second scan.
- Placebo, Then Oxytocin: Healthy adult subjects who received placebo before their first scan, and oxytocin before their second scan.
Period: MIT fMRI and MEG Resting State Study
Arm/Group | Oxytocin, Then Placebo | Placebo, Then Oxytocin
Started | 11 | 10
Completed | 10 (Enrollment completed in March 2014.) | 9
Not Completed | 1 | 1
Period: MGH Rest + Nueroeconomic Task fMRI
Arm/Group | Oxytocin, Then Placebo | Placebo, Then Oxytocin
Started | 10 (Subjects who dropped out/were excluded (10), did so before they received either Oxytocin or Placebo.) | 10
Completed | 10 (Enrollment completed in May 2015.) | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes only subjects who completed the study; i.e., received both oxytocin and placebo (19 at MIT and 20 at MGH).
Groups:
- Oxytocin, Then Placebo: Healthy adult subjects received several puffs of Syntocinon Nasal Spray, 40IU, once, prior to MRI and/or MEG scanning.
  This group contains subjects who received oxytocin prior to first scan and placebo prior to second scan.
- Placebo, Then Oxytocin: Healthy adult subjects received several puffs of Syntocinon Placebo Formulation, 40IU, once, prior to MRI and/or MEG scanning.
  This group contains subjects who received placebo prior to first scan and oxytocin prior to second scan.
- Total: Total of all reporting groups
Arm/Group | Oxytocin, Then Placebo | Placebo, Then Oxytocin | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 39
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (6.3) | 28.1 (6.9) | 27.6 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 20 | 19 | 39
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Benevolent Rounds
Description: This study recruited healthy adults. Subjects participated in an interactive neuroeconomic game, an iterative version of the classical "Trust Study." During this game, the subject ('investor') is first provided a sum of money (20 units). He then has the choice in terms of how much to invest in a fictional computer-generated trustee. The trustee then sends some percentage back to the subject ('investor'), and the game iterates over 20 trials (rounds). We computed the investment ratio as the ratio of the actual investment and the maximum allowed amount of 20 units, and analogously for the repayment ratio. Benevolent rounds were defined as those with increased investment ratios even after a decreased repayment ratio.
Time Frame: Immediately after completion of the study, for each subject.
Population: Healthy adult men.
Measure: Mean (Standard Deviation); unit: number of rounds
Groups:
- Oxytocin: Subjects received oxytocin prior to the scan.
- Placebo: Subjects received placebo prior to the scan.
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 17 | 17
number of rounds | 6.8 (2.0) | 6.8 (2.3)

2. Primary Outcome: Number of Malevolent Rounds
Description: This study recruited healthy adults. Subjects participated in an interactive neuroeconomic game, an iterative version of the classical "Trust Study." During this game, the subject ('investor') is first provided a sum of money (20 units). He then has the choice in terms of how much to invest in a fictional computer-generated trustee. The trustee then sends some percentage back to the subject ('investor'), and the game iterates over 20 trials (rounds). We computed the investment ratio as the ratio of the actual investment and the maximum allowed amount of 20 units, and analogously for the repayment ratio. Malevolent rounds were defined as those with decreased investment ratios even after an increased repayment ratio.
Time Frame: Immediately after completion of the study, for each subject.
Population: Healthy adult men.
Measure: Mean (Standard Deviation); unit: number of rounds
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 17 | 17
number of rounds | 2.8 (1.5) | 3.0 (2.1)

3. Secondary Outcome: Functional Connectivity Between OFC and AMY
Description: During functional scans, subjects participated in an interactive neuroeconomic game, an iterative version of the classical "Trust Study." Subjects participated in an interactive neuroeconomic game, an iterative version of the classical "Trust Study." During this game, the subject ('investor') is first provided a sum of money (20 units). He then has the choice in terms of how much to invest in a fictional computer-generated trustee. The trustee then sends some percentage back to the subject ('investor'), and the game iterates over 20 trials (rounds).
  Using Dynamical Causal Modeling (DCM) we modeled the dynamic interaction between amygdala (AMY), nucleus accumbens (NAcc) and the orbitofrontal cortex (OFC). We observed altered connectivity strength between AMY and OFC under OT as compared to PL conditions.
Time Frame: Within two weeks of enrollment completion.
Population: Healthy adult men (17 subjects completed the task fMRI (Trust Study) at MGH, remaining 3 subjects at MGH did not complete the task). The values reported for connections strengths below (0.45 and 0.18) are from the Bayesian Parameter Averaging. The measure of precision is the associated posterior probability, which is 1 for both.
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 17 | 17
Hz | 0.45 (NA) — The value reported for connections strength (0.45 ) is from the Bayesian Parameter Averaging. The measure of precision is the associated posterior probability, which, in this case, is 1. | 0.18 (NA) — The value reported for connections strength (0.18) is from the Bayesian Parameter Averaging. The measure of precision is the associated posterior probability, which, in this case, is 1.

ADVERSE EVENTS:
Groups:
- Oxytocin, Then Placebo: Subjects who received oxytocin before their first scan, and placebo before their second scan.
- Placebo, Then Oxytocin: Subjects who received placebo before their first scan, and oxytocin before their second scan.
Arm/Group | Oxytocin, Then Placebo | Placebo, Then Oxytocin
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

LIMITATIONS AND CAVEATS:
Data collection has been completed, but data analysis is ongoing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No